CLINICAL TRIAL: NCT01001715
Title: Randomized, Double-blind, Placebo-controlled Study of the Effect of a Single Injection of SAR164877 (REGN475) on Reduction of Pain From Vertebral Fracture Associated With Osteoporosis
Brief Title: Single Injection of REGN475/SAR164877 in Treatment of Vertebral Fracture Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision due to low subject recruitment and enrollment
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT11308
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REGN475/SAR164877 (Experimental): REGN475/SAR164877, single injection, dose depending on the participant's body weight
  Interventions: Drug: REGN475/SAR164877
- Placebo (Placebo Comparator): Placebo (for REGN475/SAR164877), single injection
  Interventions: Drug: Placebo (for REGN475/SAR164877)

INTERVENTIONS:
Drug: REGN475/SAR164877 — Pharmaceutical form: solution
  Route of administration: intravenous infusion over 30 minutes
  Arms: REGN475/SAR164877
Drug: Placebo (for REGN475/SAR164877) — Pharmaceutical form: solution
  Route of administration: intravenous infusion over 30 minutes
  Arms: Placebo

SUMMARY:
Primary objective was to demonstrate the activity of REGN475/SAR164877 in reducing the pain associated with vertebral fracture.

Secondary objectives were:

* to assess the safety and tolerability of REGN475/SAR164877 in patients with vertebral fracture pain;
* to characterize the pharmacokinetic and immunogenicity profiles of REGN475/SAR164877 in this population.

DETAILED DESCRIPTION:
The duration of the study period for each participant was up to 13 weeks, including a screening period up to 5 days, and 12-week follow-up after the injection.

ELIGIBILITY:
Inclusion criteria:

- Moderate to severe pain due to non-traumatic vertebral fracture associated with osteoporosis.

Exclusion criteria:

* Mild pain score on the Pain Intensity-Numeric Rating Scale [PI-NRS] at screening and randomization visits;
* Narcotic addiction;
* Post-fracture vertebral instability;
* Unwillingness to use study-defined rescue analgesia exclusively.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in pain intensity as assessed by Pain Intensity Numeric Rating Scale [PI-NRS] | baseline and 4 weeks after injection
  The baseline value was defined as the average of PI-NRS values obtained at screening and at randomization visit.
  The Week 4 value was defined as the average of PI-NRS values obtained daily through e-Diary assessments during Week 4.

SECONDARY OUTCOMES:
Mean change from baseline in pain intensity as assessed by PI-NRS | baseline and every other weeks up to 12 weeks after injection
Percentage of pain-free days (score "0" pain on PI-NRS) | 12 weeks
Percentage of days with rescue analgesia use | 12 weeks
Change from baseline in Quality of Life Questionnaire of the European Foundation for Osteoporosis [QUALEFFO] score | baseline and 4, 8, 12 weeks
Change from baseline in Short Form-12 Item Quality of Life Questionnaire [SF-12] score | baseline and 4, 8, 12 weeks
Patient Global Impression of Change [PGIC] score | 4, 8, 12 weeks
Percentage of participants with at least 30% and 50% reduction from baseline in pain intensity | up to 12 weeks after injection
Pharmacokinetic: REGN475/SAR164877 serum concentration | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- United States (11):
  - Sanofi-Aventis Investigational Site Number 840005, Beverly Hills, California
  - Sanofi-Aventis Investigational Site Number 840001, Fresno, California
  - Sanofi-Aventis Investigational Site Number 840017, Sacramento, California
  - Sanofi-Aventis Investigational Site Number 840028, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840008, Stockton, California
  - Sanofi-Aventis Investigational Site Number 840013, Boynton Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840047, Clearwater, Florida
  - Sanofi-Aventis Investigational Site Number 840034, Atlanta, Georgia
  - Sanofi-Aventis Investigational Site Number 840026, New York, New York
  - Sanofi-Aventis Investigational Site Number 840044, Fort Worth, Texas
  - Sanofi-Aventis Investigational Site Number 840023, Southlake, Texas